CLINICAL TRIAL: NCT03324568
Title: Helping Young Children Improve Eating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kelly Tanner (Other)
Responsible Party: Sponsor-Investigator, Kelly Tanner, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB17-00420
Record Dates: First submitted 2017-10-17; First posted 2017-10-27 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Feeding and Eating Disorders of Childhood
MeSH Terms: conditions — Feeding and Eating Disorders of Childhood

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational handout (Other)
  Interventions: Behavioral: Educational Handout
- Video plus educational handout (Experimental)
  Interventions: Behavioral: Parent Education Videos; Behavioral: Educational Handout

INTERVENTIONS:
Behavioral: Parent Education Videos — Participants will receive educational videos describing behavioral techniques to improve parent and child eating behavior.
  Arms: Video plus educational handout
Behavioral: Educational Handout — Participants will receive educational handouts describing behavioral techniques to improve parent and child eating behavior.

SUMMARY:
This study will evaluate the impact of different types of educational materials on parent and child feeding behaviors. Specifically, the investigators will test the feasibility, acceptability, and effectiveness of an investigator-developed series of parent training videos designed to teach behavioral strategies to promote feeding in young children with feeding difficulties.

ELIGIBILITY:
Inclusion Criteria:

* Parents of patients ages 18 months through 6 years currently on the waitlist (for an estimated time of at least 4-6 weeks) for outpatient feeding therapy, or with feeding concerns identified in a primary care visit; English-speaking parents; parent has the technology to access the videos and REDCap survey.

Exclusion Criteria:

* Parents of patients not currently eating by mouth; parents of patients currently being treated by a psychologist, occupational therapist, or speech therapist to address feeding, eating, or swallowing skills; parents of patients who have aspirated on their most recent videofluoroscopic swallow study or who currently have a tracheostomy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2018-02-04 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
Behavioral Pediatrics Feeding Assessment | 4 weeks
  Parent questionnaire that measures parent and child feeding behaviors and attitudes. A higher score indicates more difficulties.

SECONDARY OUTCOMES:
Food Frequency Questionnaire | 4 weeks
  Parent questionnaire that measures the amount of different foods children ate over a specific time period (e.g. one month). A higher score indicates more different foods were consumed by the child.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided
Not yet decided.